CLINICAL TRIAL: NCT02125123
Title: Oral Nutritional Supplementation in Children With Picky Eating Behaviors
Brief Title: Oral Nutritional Supplementation in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AL15
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Children
MeSH Terms: interventions — Dietary Supplements; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional Supplement and Counseling (Experimental): Two servings a day; ready-to-feed nutritional supplement plus dietary counseling
  Interventions: Other: Nutritional Supplement and Counseling
- Counseling (Active Comparator): Dietary Counseling
  Interventions: Other: Counseling

INTERVENTIONS:
Other: Nutritional Supplement and Counseling — Ready-to-feed nutritional supplement and dietary counseling
  Arms: Nutritional Supplement and Counseling
Other: Counseling — Dietary counseling
  Arms: Counseling

SUMMARY:
This study will investigate the effect of an oral nutritional supplement (ONS) along with dietary counseling on improving the dietary intake among children with picky eating behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 36 months and < 109 months of age.
2. Healthy and not suffering from any physical disability.
3. Height-for-age and BMI-for-age between the 5th and the 95th percentile; weight-for-age between the 5th and the 85th percentile.
4. Capable of oral feeding.
5. Has a mean score of greater than 3.0 on the fussiness category in the Children's Eating Behaviour Questionnaire and also consumes on average less than the daily recommendations for at least 3 of 5 food groups (Dietary Guidelines for America, 2010).
6. Willing to abstain from consuming non-study nutritional supplements during the study intervention period.

Exclusion Criteria:

1. History of an acute or chronic condition that may affect feeding habits or nutritional status.
2. Taking any medications or nutritional supplements on a daily basis for more than 2 weeks during the past month that may profoundly affect feeding habits or nutritional status.
3. Clinically significant nutritional deficiency requiring specific treatment with any other nutritional supplement.
4. Any acute/chronic condition requiring medical treatment which may include hospitalization.
5. Allergy or intolerance to any ingredient in the study product.
6. Gastrointestinal infection, acute constipation or acute diarrhea.
7. Hepatitis B or C, or HIV, or malignancy.
8. Congenital cardiac defects.
9. Dysphagia, aspiration risk or difficulty in swallowing due to acquired/congenital abnormalities.
10. Parent(s)/LG of the subject has any clinically significant medical disease or physical/psychological condition that may interfere with protocol adherence or ability of the parent(s)/LG to give informed consent.

Ages: 36 Months to 109 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Vitamin D Intake | Change from Baseline to Week 4

SECONDARY OUTCOMES:
Macronutrient Intake | Change from Baseline to Week 4
  24-hour dietary recall interview
Micronutrient Intake | Change from Baseline to Week 4
  24-hour dietary recall interview

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Williams, MPH, Study Chair — Abbott Nutrition
Locations (2):
- United States (2):
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Radiant Research, Inc., Cincinnati, Ohio